CLINICAL TRIAL: NCT04607447
Title: Effectiveness and Safety of Low Intracranial Pressure Treatment Strategies for Patients With Chronic Subdural Hematoma - A Randomized, Controlled, Multi-center Clinical Study
Brief Title: Low Intracranial Pressure Treatment Strategies for Chronic Subdural Hematoma Patients
Acronym: CSDH-LP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xuehai Wu, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2020-063
Record Dates: First submitted 2020-10-26; First posted 2020-10-29 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Chronic Subdural Hematoma
Keywords: Low intracranial pressure
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Intracranial Hypotension | interventions — Atorvastatin; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin plus Dexamethasone tablets (Active Comparator)
  Interventions: Drug: Atorvastatin plus Dexamethasone
- drugs+low intracranial pressure strategy treatment (Experimental): Drugs means treatment with Atorvastatin plus Dexamethasone tablets
  Interventions: Behavioral: low intracranial pressure strategy treatment; Drug: Atorvastatin plus Dexamethasone

INTERVENTIONS:
Behavioral: low intracranial pressure strategy treatment — 1. Supine position for 16h-18h daily, with head toward the affected side in most of the time, and 15-20 cm elevation of lower limbs.
  2. Abdominal belt compression
  Arms: drugs+low intracranial pressure strategy treatment
Drug: Atorvastatin plus Dexamethasone — Atorvastatin plus Dexamethasone

SUMMARY:
The proportion of the elderly population is increasing rapidly. Chronic subdural hematoma has become the most common cause of surgery in neurosurgery for elderly patients. The standard treatment for cSDH is mostly surgery. Clinically, we often encounter elderly patients with certain underlying diseases or organ dysfunction, especially preexisting cardiovascular disease or medication history like anticoagulant or antiplatelet drugs, resulting in poor surgical tolerance, high risk during anesthesia and hematoma recurrence. At present, the mechanism of cSDH is not completely clear. Our previous observational studies had shown significant correlation between cSDH and intracranial hypotension. So we would like to conduct a randomized, controlled, multi-center clinical study to explore the effectiveness and safety of low intracranial pressure treatment strategies for patients with chronic subdural hematoma.

ELIGIBILITY:
Inclusion Criteria:

* patients above 14 yrs with chronic subdural hematoma confirmed by cranial imaging;
* patients with MGS-GCS score ≤1 point, showing no signs of neurological deficits caused by CSDH or characteristics of high intracranial pressure;
* patients with MGS-GCS score ≥1 point, but with medication history of anticoagulant or antiplatelet drugs, coagulation dysfunction so that they are unsuitable or intolerant of surgery although they are in stable condition;
* patients who are unwilling to operate when they have no life-threatening brain herniation or no indications for emergency surgery, which confirmed by two neurosurgeons

Exclusion Criteria:

* women pregnant or in lactation
* those who are allergic to atorvastatin, hypoxamethasone;
* patients with brain herniation or altered mental status;
* patients with primary diseases like tumors, hemorrhagic diseases or some other critically serious conditions( eg.multiple organ failure);
* patients with uncontrollable diabetes and heart failure
* patients with preexisting chronic abdominal diseases (such as inflammatory bowel disease) or lung tumors or digestive system neoplasm
* Patients with abnormal liver function
* patients had taken atorvastatin or dexamethasone, ACEI in the past one week
* other conditions not eligible to enroll the trial confirmed by two individual doctor

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
subdural hematoma volume | three months
  difference of hematoma volume in subdura between two groups
Markwalder scale | three months
  difference of Markwalder scale between two groups;The Markwalder Scale is designed to measure the chronic subdural hematoma scale. This scale is categorized into four grade. Grade 0 denots the patient neurologically normal, whereas grade 4, the highest grade, denotes the worst neuological assessment.
Modified Rankin Scale | three months
  difference of Modified Rankin Scale between two groups; The modified Rankin Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death.
Extended Glasgow Outcome score | three months
  difference of Extended Glasgow Outcome score between two groups; This score is used to measure the outcome after neurological disease. It defines 5 categories of possible outcomes after a brain injury, which is from good recovery(5) to death(1).

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No